CLINICAL TRIAL: NCT06777043
Title: Long-term Remission After Ileorectal Anastomosis in Crohn's Disease.
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: IRA
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: IBD - Inflammatory Bowel Disease
Keywords: IBD; CD; IRA
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with isolated colonic Crohn's disease: The first group had isolated colonic Crohn's disease without rectal involvement and perianal disease
- Patients with rectal and/or ileal Crohn's disease: the second group included patients who had rectal and/or ileal involvement, with or without perianal disease

SUMMARY:
Single-center, retrospective, observational study. The medical records of patients who underwent colectomy and ileorectal anastomosis (IRA) for refractory Crohn's colitis between 1996 and 2016 were reviewed.

DETAILED DESCRIPTION:
Several studies show that, although the type of disease changes in a statistically significant way after 5 years from diagnosis, overall, a follow-up of more than 10 years indicates that the disease remains unchanged in about 85% of patients. Studies show that up to 70% of patients with Crohn's disease (CD) undergo surgery at least once in their lifetime. In colon Crohn's disease, the cumulative risk of surgery 10 years after diagnosis is lower compared to ileal Crohn's disease. For patients with extensive colitis who do not respond to medical therapy, total colectomy with ileorectal anastomosis (IRA) is a safe and effective approach. Several studies in the literature have retrospectively evaluated the recurrence rate after colectomy and IRA in Crohn's disease-related colitis, showing reasonable recurrence rates. Furthermore, several studies have highlighted that rectal involvement and the presence of perianal disease may be predictive factors for recurrence in Crohn's colitis treated with colectomy and ileorectal anastomosis (IRA). Ileal involvement in colectomy in patients with Crohn's colitis appears to be associated with a higher risk of recurrence in the small intestine and failure of the IRA. Our study is based on the hypothesis that, in patients with extensive and refractory Crohn's colitis but without rectal involvement or perianal disease, colectomy and IRA could instead drastically reduce the recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* patients with Crohn's colitis who underwent colectomy and ileorectal anastomosis

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Crohn's disease who underwent colectomy and ileorectal anastomosis between 1996 and 2016, in a single IBD tertiary center
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Recurrence of disease | within 2 years of the surgery
  Recurrence of disease

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rizzello, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

REFERENCES:
- [Background] Salice M, Rizzello F, Sgambato D, Calabrese C, Manguso F, Laureti S, Rottoli M, Poggioli G, Gionchetti P. Long term remission after ileorectal anastomosis in Crohn's colitis. Dig Liver Dis. 2021 May;53(5):592-597. doi: 10.1016/j.dld.2020.06.021. Epub 2020 Jun 29. PMID 32616463
- See also: "Long term remission after ileorectal anastomosis in Crohn's colitis" — https://pubmed.ncbi.nlm.nih.gov/32616463/